CLINICAL TRIAL: NCT00005145
Title: Study of Trends in Cardiovascular Risk Factors in an Urban Population.
Brief Title: Minnesota Heart Survey - Risk Factor Survey
Acronym: MHS
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1016; R01HL023727 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Cerebrovascular Accident; Coronary Disease; Hypertension; Myocardial Infarction
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Stroke; Coronary Disease; Hypertension; Myocardial Infarction

GROUPS / COHORTS (1):
- Observational, no interventions

SUMMARY:
To continue surveillance of cardiovascular disease risk factors in the seven-county area of Minneapolis-St. Paul.

DETAILED DESCRIPTION:
BACKGROUND:

Cardiovascular disease mortality rates, especially for myocardial infarction and stroke, have fallen markedly over the past several decades in all race, sex, and age groups in the United States. Between 1966 and 1986, the combined death rate for all cardiovascular diseases declined by 42 percent. In 1986, the death rate for coronary heart disease was 55 percent of what it had been in 1966, and cerebrovascular disease was 42 percent of what it had been in 1966. The decline is assumed to be related to several factors including improved medical care and risk factor modification for elevated blood lipids, cigarette smoking, and hypertension. The Minnesota Heart Survey provide trends (1970-2002) in coronary heart disease deaths out-of-hospital, in hospitalization rates, case fatality and survivorship for myocardial infarction and stroke in the metropolitan area.

DESIGN NARRATIVE:

Between 1979 and 1999, R01HL23727 supported mortality surveillance and morbidity surveillance. Beginning in FY 2000, R01HL65755 supports the morbidity and mortality surveillance and R01HL23727 supports the risk factor survey.

Mortality Surveillance: The mortality surveillance was a continuation of a surveillance study performed by the investigators since 1960 for the state of Minnesota. Mortality data for hypertension, stroke, coronary heart disease, and all cardiovascular renal disease were monitored for the Twin City metropolitan area with a total population of two million. Age, sex, area, location of death and cause-specific death rates were followed. Trends in cancer, diabetes, and other non-cardiovascular disease were examined. Case fatality rates, including one- and five-year survivorships were determined and related to coronary heart disease mortality trends.

Morbidity Surveillance: All discharges from the seven-county area hospitals with acute and chronic myocardial heart disease and stroke listed among the discharge diagnoses were recorded using Professional Standards Review Organization data tapes. A ten percent random sample of all recorded diagnoses were validated yearly by abstracting data from hospital records. Each year's validation sample of definite and probable cases of myocardial infarction and stroke formed a cohort to be followed for mortality for one year after the onset of the disease event. Individual hospitals and the Professional Standards Review Organization in the area provided data on the total numbers of coronary care unit admissions and coronary artery bypass operations for each year. Beginning in August 1988, a registry was established for all new incident cases of coronary heart disease at the University of Minnesota Hospital and the Ramsey County Hospital. In 1989, twelve hospitals were part of the myocardial infarction registry.

Risk Factor Surveillance: Population samples, aged 25-74 years, are recruited and measured for blood pressure, serum cholesterol, serum high density lipoprotein cholesterol, cigarette smoking, diet, physical activity, height, weight, health attitudes and beliefs, and coronary prone behavior. Surveys were completed in 1980-1982 and 1984-1985. The third survey conducted in 1990-1992 included the Willett Food Frequency Questionnaire and bioimpedance measurements. A nested case-control study using the 1980-1982 risk factor cohort examined the baseline cardiovascular disease risk factor differences between coronary heart disease in cases and controls.

The study was renewed in the year 2000 under R01HL23727 to conduct a population survey of 4,000 adults, ages 25 to 84 in 2000-2002, to detect current trends in cardiovascular disease risk factors, including serum lipids, blood pressure, cigarette smoking prevalence, dietary fat intake, obesity, diabetes, physical inactivity, fibrinogen, and serum vitamin E. Cohort and ecological analyses will be used to link secular trends in risk factors to morbidity and mortality from coronary heart disease, congestive heart failure, and stroke. A total of 1,000 children and adolescents, ages 8-17, will also be surveyed using youth-specific measurement instruments where appropriate.

ELIGIBILITY:
No eligibility criteria

Ages: 8 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1979-04; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Cardiovascular risk factor trends | 26 years

CONTACTS AND LOCATIONS:
Overall Officials: Donna Arnett — University of Minnesota

REFERENCES:
- [Background] Luepker RV, Rastam L, Hannan PJ, Murray DM, Gray C, Baker WL, Crow R, Jacobs DR Jr, Pirie PL, Mascioli SR, Mittelmark MB, Blackburn H. Community education for cardiovascular disease prevention. Morbidity and mortality results from the Minnesota Heart Health Program. Am J Epidemiol. 1996 Aug 15;144(4):351-62. doi: 10.1093/oxfordjournals.aje.a008936. PMID 8712192
- [Background] Rosamond WD, Shahar E, Luepker RV. Assessing medical history in coronary heart disease surveillance: agreement between contemporaneous and retrospective methods. Epidemiology. 1996 Jul;7(4):447-9. doi: 10.1097/00001648-199607000-00020. PMID 8793376
- [Background] Pieper RM, Arnett DK, McGovern PG, Shahar E, Blackburn H, Luepker RV. Trends in cholesterol knowledge and screening and hypercholesterolemia awareness and treatment, 1980-1992. The Minnesota Heart Survey. Arch Intern Med. 1997 Nov 10;157(20):2326-32. PMID 9361573
- [Background] McGovern PG, Herlitz J, Pankow JS, Karlsson T, Dellborg M, Shahar E, Luepker RV. Comparison of medical care and one- and 12-month mortality of hospitalized patients with acute myocardial infarction in Minneapolis-St. Paul, Minnesota, United States of America and Goteborg, Sweden. Am J Cardiol. 1997 Sep 1;80(5):557-62. doi: 10.1016/s0002-9149(97)00421-9. PMID 9294981
- [Background] Iribarren C, Luepker RV, McGovern PG, Arnett DK, Blackburn H. Twelve-year trends in cardiovascular disease risk factors in the Minnesota Heart Survey. Are socioeconomic differences widening? Arch Intern Med. 1997 Apr 28;157(8):873-81. PMID 9129547
- [Background] Shahar E, Lewis M, Keil U, McGovern PG, Lowel H, Luepker RV. Hospital care and survival of acute myocardial infarction patients in Minnesota and southern Germany: a comparative study. Coron Artery Dis. 1996 Jun;7(6):467-73. doi: 10.1097/00019501-199606000-00010. PMID 8889363
- [Background] Venters MH, Jacobs DR Jr, Luepker RV, Maiman LA, Gillum RF. Spouse concordance of smoking patterns: the Minnesota Heart Survey. Am J Epidemiol. 1984 Oct;120(4):608-16. doi: 10.1093/oxfordjournals.aje.a113922. PMID 6475929
- [Background] Gillum RF, Liu KC. Coronary heart disease mortality in United States blacks, 1940-1978: trends and unanswered questions. Am Heart J. 1984 Sep;108(3 Pt 2):728-32. doi: 10.1016/0002-8703(84)90665-3. No abstract available. PMID 6475741
- [Background] Folsom AR, Prineas RJ, Jacobs DR, Luepker RV, Gillum RF. Measured differences between fourth and fifth phase diastolic blood pressures in 4885 adults: implications for blood pressure surveys. Int J Epidemiol. 1984 Dec;13(4):436-41. doi: 10.1093/ije/13.4.436. PMID 6519881
- [Background] Folsom AR, Caspersen CJ, Taylor HL, Jacobs DR Jr, Luepker RV, Gomez-Marin O, Gillum RF, Blackburn H. Leisure time physical activity and its relationship to coronary risk factors in a population-based sample. The Minnesota Heart Survey. Am J Epidemiol. 1985 Apr;121(4):570-9. doi: 10.1093/oxfordjournals.aje.a114035. PMID 4014146
- [Background] Gillum RF, Gomez-Marin O, Kottke TE, Jacobs DR Jr, Prineas RJ, Folsom AR, Luepker RV, Blackburn H. Acute stroke in a metropolitan area, 1970 and 1980. The Minnesota Heart Survey. J Chronic Dis. 1985;38(11):891-8. doi: 10.1016/0021-9681(85)90124-9. PMID 4055977
- [Background] Luepker RV, Jacobs DR, Gillum RF, Folsom AR, Prineas RJ, Blackburn H. Population risk of cardiovascular disease: the Minnesota Heart Survey. J Chronic Dis. 1985;38(8):671-82. doi: 10.1016/0021-9681(85)90021-9. PMID 4019704
- [Background] Pechacek TF, Folsom AR, de Gaudermaris R, Jacobs DR Jr, Luepker RV, Gillum RF, Blackburn H. Smoke exposure in pipe and cigar smokers. Serum thiocyanate measures. JAMA. 1985 Dec 20;254(23):3330-2. PMID 4068167
- [Background] Sorensen G, Pirie P, Folsom A, Luepker R, Jacobs D, Gillum R. Sex differences in the relationship between work and health: the Minnesota Heart Survey. J Health Soc Behav. 1985 Dec;26(4):379-94. No abstract available. PMID 4086760
- [Background] Folsom AR, Smith CL, Prineas RJ, Grimm RH Jr. Serum calcium fractions in essential hypertensive and matched normotensive subjects. Hypertension. 1986 Jan;8(1):11-5. doi: 10.1161/01.hyp.8.1.11. PMID 3943882
- [Background] Venters M, Jacobs DR Jr, Pirie P, Luepker RV, Folsom AR, Gillum RF. Marital status and cardiovascular risk: the Minnesota Heart Survey and the Minnesota Heart Health Program. Prev Med. 1986 Nov;15(6):591-605. doi: 10.1016/0091-7435(86)90064-2. PMID 3797391
- [Background] Folsom AR, Jacobs DR Jr, Caspersen CJ, Gomez-Marin O, Knudsen J. Test-retest reliability of the Minnesota Leisure Time Physical Activity Questionnaire. J Chronic Dis. 1986;39(7):505-11. doi: 10.1016/0021-9681(86)90195-5. PMID 3722314
- [Background] Folsom AR, Jacobs DR, Luepker RV, Kushi LH, Gillum RF, Elmer PJ, Blackburn H. Nutrient intake in a metropolitan area, 1973-74 vs 1980-82: the Minnesota Heart Survey. Am J Clin Nutr. 1987 Jun;45(6):1533-40. doi: 10.1093/ajcn/45.6.1533. PMID 3591733
- [Background] Gomez-Marin O, Folsom AR, Kottke TE, Wu SC, Jacobs DR Jr, Gillum RF, Edlavitch SA, Blackburn H. Improvement in long-term survival among patients hospitalized with acute myocardial infarction, 1970 to 1980. The Minnesota Heart Survey. N Engl J Med. 1987 May 28;316(22):1353-9. doi: 10.1056/NEJM198705283162201. PMID 3574412
- [Background] Folsom AR, Gomez-Marin O, Gillum RF, Kottke TE, Lohman W, Jacobs DR Jr. Out-of-hospital coronary death in an urban population--validation of death certificate diagnosis. The Minnesota Heart Survey. Am J Epidemiol. 1987 Jun;125(6):1012-8. doi: 10.1093/oxfordjournals.aje.a114617. PMID 3578243
- [Background] Folsom AR, Gomez-Marin O, Sprafka JM, Prineas RJ, Edlavitch SA, Gillum RF. Trends in cardiovascular risk factors in an urban black population, 1973-74 to 1985: the Minnesota Heart Survey. Am Heart J. 1987 Nov;114(5):1199-205. doi: 10.1016/0002-8703(87)90197-9. PMID 3673887
- [Background] Hahn LP, Folsom AR, Sprafka JM, Prineas RJ. Prevalence and accuracy of home sphygmomanometers in an urban population. Am J Public Health. 1987 Nov;77(11):1459-61. doi: 10.2105/ajph.77.11.1459. PMID 3661803
- [Background] Sorensen G, Jacobs DR Jr, Pirie P, Folsom A, Luepker R, Gillum R. Relationships among type A behavior, employment experiences, and gender: the Minnesota Heart Survey. J Behav Med. 1987 Aug;10(4):323-36. doi: 10.1007/BF00846473. PMID 3669068
- [Background] Burke GL, Folsom AR, Crow RS, Edlavitch SE, Sprafka JM: Validating Death Certificate Diagnosis of Coronary Heart Disease Using Community Data Sources. Proceedings of Public Health Conference on Records and Statistics, DHHS Pub. No(PHS) 88-1214:179-182, 1988
- [Background] Edlavitch SA, Baxter J. Comparability of mortality follow-up before and after the National Death Index. Am J Epidemiol. 1988 Jun;127(6):1164-78. doi: 10.1093/oxfordjournals.aje.a114910. PMID 3369416
- [Background] Folsom AR, Iso H, Sprafka JM, Edlavitch SA, Luepker RV. Use of aspirin for prevention of cardiovascular disease--1981-82 to 1985-86: the Minnesota Heart Survey. Am Heart J. 1988 Sep;116(3):827-30. doi: 10.1016/0002-8703(88)90344-4. PMID 3261930
- [Background] Luepker RV, Jacobs DR Jr, Folsom AR, Gillum RF, Frantz ID Jr, Gomez O, Blackburn H. Cardiovascular risk factor change--1973-74 to 1980-82: the Minnesota Heart Survey. J Clin Epidemiol. 1988;41(9):825-33. doi: 10.1016/0895-4356(88)90098-4. PMID 3183688
- [Background] Kushi LH, Folsom AR, Jacobs DR Jr, Luepker RV, Elmer PJ, Blackburn H. Educational attainment and nutrient consumption patterns: the Minnesota Heart Survey. J Am Diet Assoc. 1988 Oct;88(10):1230-6. PMID 2844877
- [Background] Sprafka JM, Folsom AR, Burke GL, Edlavitch SA. Prevalence of cardiovascular disease risk factors in blacks and whites: the Minnesota Heart Survey. Am J Public Health. 1988 Dec;78(12):1546-9. doi: 10.2105/ajph.78.12.1546. PMID 3263810
- [Background] Sprafka JM, Folsom AR, Burke GL, Edlavitch SA. Prevalence of coronary heart disease risk factors in an urban black population: the Minnesota Heart Survey, 1985. Prev Med. 1988 May;17(3):321-34. doi: 10.1016/0091-7435(88)90007-2. PMID 3405987
- [Background] Folsom AR, Sprafka JM, Luepker RV, Jacobs DR Jr. Beliefs among black and white adults about causes and prevention of cardiovascular disease: the Minnesota Heart Survey. Am J Prev Med. 1988 May-Jun;4(3):121-7. PMID 3395497
- [Background] Burke GL, Edlavitch SA, Crow RS. The effects of diagnostic criteria on trends in coronary heart disease morbidity: the Minnesota Heart Survey. J Clin Epidemiol. 1989;42(1):17-24. doi: 10.1016/0895-4356(89)90021-8. PMID 2643674
- [Background] Mascioli SR, Jacobs DR Jr, Kottke TE. Diagnostic criteria for hospitalized acute myocardial infarction: the Minnesota experience. Int J Epidemiol. 1989 Mar;18(1):76-83. doi: 10.1093/ije/18.1.76. PMID 2656562
- [Background] Burke GL, Sprafka JM, Folsom AR, Luepker RV, Norsted SW, Blackburn H. Trends in CHD mortality, morbidity and risk factor levels from 1960 to 1986: the Minnesota Heart Survey. Int J Epidemiol. 1989;18(3 Suppl 1):S73-81. PMID 2807710
- [Background] Sprafka JM, Burke GL, Folsom AR, Hahn LP. Hypercholesterolemia prevalence, awareness, and treatment in blacks and whites: the Minnesota Heart Survey. Prev Med. 1989 Jul;18(4):423-32. doi: 10.1016/0091-7435(89)90002-9. PMID 2798366
- [Background] Edlavitch SA, Crow R, Burke GL, Huber J, Prineas R, Blackburn H. The effect of the number of electrocardiograms analyzed on cardiovascular disease surveillance: the Minnesota Heart Survey (MHS). J Clin Epidemiol. 1990;43(1):93-9. doi: 10.1016/0895-4356(90)90061-s. PMID 2319286
- [Background] Sprafka JM, Burke GL, Folsom AR, Luepker RV, Blackburn H. Continued decline in cardiovascular disease risk factors: results of the Minnesota Heart Survey, 1980-1982 and 1985-1987. Am J Epidemiol. 1990 Sep;132(3):489-500. doi: 10.1093/oxfordjournals.aje.a115685. PMID 2389753
- [Background] Iso H, Jacobs DR Jr, Goldman L. Accuracy of death certificate diagnosis of intracranial hemorrhage and nonhemorrhagic stroke. The Minnesota Heart Survey. Am J Epidemiol. 1990 Nov;132(5):993-8. doi: 10.1093/oxfordjournals.aje.a115742. PMID 2239914
- [Background] Lilienfeld DE, Godbold JH, Burke GL, Sprafka JM, Pham DL, Baxter J. Hospitalization and case fatality for pulmonary embolism in the twin cities: 1979-1984. Am Heart J. 1990 Aug;120(2):392-5. doi: 10.1016/0002-8703(90)90085-c. PMID 2382617
- [Background] Sprafka JM, Folsom AR, Burke GL, Hahn LP, Pirie P. Type A behavior and its association with cardiovascular disease prevalence in blacks and whites: the Minnesota Heart Survey. J Behav Med. 1990 Feb;13(1):1-13. doi: 10.1007/BF00844896. PMID 2348446
- [Background] Demirovic J, Sprafka JM, Folsom AR, Laitinen D, Blackburn H. Menopause and serum cholesterol: differences between blacks and whites. The Minnesota Heart Survey. Am J Epidemiol. 1992 Jul 15;136(2):155-64. doi: 10.1093/oxfordjournals.aje.a116482. PMID 1357959
- [Background] McGovern PG, Burke GL, Sprafka JM, Xue S, Folsom AR, Blackburn H. Trends in mortality, morbidity, and risk factor levels for stroke from 1960 through 1990. The Minnesota Heart Survey. JAMA. 1992 Aug 12;268(6):753-9. PMID 1640576
- [Background] Naughton MJ, Luepker RV, Sprafka JM, McGovern PG, Burke GL. Community trends in CPR training and use: the Minnesota Heart Survey. Ann Emerg Med. 1992 Jun;21(6):698-703. doi: 10.1016/s0196-0644(05)82782-9. PMID 1590610
- [Background] Folsom AR, Cook TC, Sprafka JM, Burke GL, Norsted SW, Jacobs DR Jr. Differences in leisure-time physical activity levels between blacks and whites in population-based samples: the Minnesota Heart Survey. J Behav Med. 1991 Feb;14(1):1-9. doi: 10.1007/BF00844764. PMID 2038041
- [Background] Burke GL, Sprafka JM, Folsom AR, Hahn LP, Luepker RV, Blackburn H. Trends in serum cholesterol levels from 1980 to 1987. The Minnesota Heart Survey. N Engl J Med. 1991 Apr 4;324(14):941-6. doi: 10.1056/NEJM199104043241402. PMID 2002818
- [Background] Edlavitch SA, Crow R, Burke GL, Baxter J. Secular trends in Q wave and non-Q wave acute myocardial infarction. The Minnesota Heart Survey. Circulation. 1991 Feb;83(2):492-503. doi: 10.1161/01.cir.83.2.492. PMID 1991368
- [Background] Sprafka JM, Norsted SW, Folsom AR, Burke GL, Luepker RV. Life-style factors do not explain racial differences in high-density lipoprotein cholesterol: the Minnesota Heart Survey. Epidemiology. 1992 Mar;3(2):156-63. doi: 10.1097/00001648-199203000-00014. PMID 1576221
- [Background] Demirovic J, Blackburn H, McGovern P, Sprafka JM, Doliszny K. Sex differences in coronary heart disease mortality trends: the Minnesota Heart Survey, 1970-1988. Epidemiology. 1993 Jan;4(1):79-82. doi: 10.1097/00001648-199301000-00015. PMID 8420587
- [Background] McGovern PG, Pankow JS, Shahar E, Doliszny KM, Folsom AR, Blackburn H, Luepker RV. Recent trends in acute coronary heart disease--mortality, morbidity, medical care, and risk factors. The Minnesota Heart Survey Investigators. N Engl J Med. 1996 Apr 4;334(14):884-90. doi: 10.1056/NEJM199604043341403. PMID 8596571
- [Background] Demirovic J, Blackburn H, McGovern PG, Luepker R, Sprafka JM, Gilbertson D. Sex differences in early mortality after acute myocardial infarction (the Minnesota Heart Survey). Am J Cardiol. 1995 Jun 1;75(16):1096-101. doi: 10.1016/s0002-9149(99)80737-1. PMID 7762492
- [Background] Rosamond WD, Sprafka JM, McGovern PG, Nelson M, Luepker RV. Validation of self-reported history of acute myocardial infarction: experience of the Minnesota Heart Survey Registry. Epidemiology. 1995 Jan;6(1):67-9. doi: 10.1097/00001648-199501000-00013. PMID 7888449
- [Background] Brodin EC, Shahar E, Rosamond WD, McGovern PG, Sprafka JM, Doliszny KM, Luepker RV. Apparently coronary heart disease-free patients in the coronary care unit: characteristics, medical care, and 1-year outcome. Coron Artery Dis. 1994 Sep;5(9):737-43. PMID 7858763
- [Background] Shahar E, McGovern PG, Sprafka JM, Pankow JS, Doliszny KM, Luepker RV, Blackburn H. Improved survival of stroke patients during the 1980s. The Minnesota Stroke Survey. Stroke. 1995 Jan;26(1):1-6. doi: 10.1161/01.str.26.1.1. PMID 7839376
- [Background] Luepker RV, Rosamond WD, Murphy R, Sprafka JM, Folsom AR, McGovern PG, Blackburn H. Socioeconomic status and coronary heart disease risk factor trends. The Minnesota Heart Survey. Circulation. 1993 Nov;88(5 Pt 1):2172-9. doi: 10.1161/01.cir.88.5.2172. PMID 8222112
- [Background] Gillum RF, Prineas RJ, Luepker RV, Taylor HL, Jacobs DR Jr, Kottke TE, Blackburn H. Decline in coronary deaths: a search for explanations. The Minnesota Mortality and Morbidity Surveillance Program. Minn Med. 1982 Apr;65(4):235-8. No abstract available. PMID 7078544
- [Background] Gillum RF, Blackburn H, Feinleib M. Current strategies for explaining the decline in ischemic heart disease mortality. J Chronic Dis. 1982;35(6):467-74. doi: 10.1016/0021-9681(82)90061-3. PMID 7076787
- [Background] Gillum RF. Coronary heart disease in black populations. I. Mortality and morbidity. Am Heart J. 1982 Oct;104(4 Pt 1):839-51. doi: 10.1016/0002-8703(82)90021-7. No abstract available. PMID 7124597
- [Background] Gillum RF, Grant CT. Coronary heart disease in black populations. II. Risk factors. Am Heart J. 1982 Oct;104(4 Pt 1):852-64. doi: 10.1016/0002-8703(82)90022-9. No abstract available. PMID 7124598
- [Background] Gillum RF, Hannan PJ, Prineas RJ, Jacobs DR Jr, Gomez-Marin O, Luepker RV, Baxter J, Kottke TE, Blackburn H. Coronary heart disease mortality trends in Minnesota, 1960-80: the Minnesota Heart Survey. Am J Public Health. 1984 Apr;74(4):360-2. doi: 10.2105/ajph.74.4.360. PMID 6703165
- [Background] Gillum RF, Folsom A, Luepker RV, Jacobs DR Jr, Kottke TE, Gomez-Marin O, Prineas RJ, Taylor HL, Blackburn H. Sudden death and acute myocardial infarction in a metropolitan area, 1970-1980. The Minnesota Heart Survey. N Engl J Med. 1983 Dec 1;309(22):1353-8. doi: 10.1056/NEJM198312013092203. PMID 6633597
- [Background] Folsom AR, Luepker RV, Gillum RF, Jacobs DR, Prineas RJ, Taylor HL, Blackburn H. Improvement in hypertension detection and control from 1973-1974 to 1980-1981. The Minnesota Heart Survey experience. JAMA. 1983 Aug 19;250(7):916-21. PMID 6345835
- [Background] Gillum RF, Fortmann SP, Prineas RJ, Kottke TE. International diagnostic criteria for acute myocardial infarction and acute stroke. Am Heart J. 1984 Jul;108(1):150-8. doi: 10.1016/0002-8703(84)90558-1. No abstract available. PMID 6731265
- [Background] Gillum RF, Jacobs DR Jr, Luepker RV, Prineas RJ, Hannan P, Baxter J, Gomez-Marin O, Kottke TE, Blackburn H. Cardiovascular mortality trends in Minnesota, 1960-1978. The Minnesota Heart Survey. J Chronic Dis. 1984;37(4):301-9. doi: 10.1016/0021-9681(84)90138-3. PMID 6715496
- [Background] Murphy RJ, Luepker RV, Jacobs DR Jr, Gillum RF, Folsom AR, Blackburn H. Citizen cardiopulmonary resuscitation training and use in a metropolitan area: the Minnesota Heart Survey. Am J Public Health. 1984 May;74(5):513-5. doi: 10.2105/ajph.74.5.513. PMID 6711735
- [Background] Folsom AR, Pechacek TF, de Gaudemaris R, Luepker RV, Jacobs DR Jr, Gillum RF. Consumption of 'low-yield' cigarettes: its frequency and relationship to serum thiocyanate. Am J Public Health. 1984 Jun;74(6):564-8. doi: 10.2105/ajph.74.6.564. PMID 6426329
- [Background] Jeffery RW, Folsom AR, Luepker RV, Jacobs DR Jr, Gillum RF, Taylor HL, Blackburn H. Prevalence of overweight and weight loss behavior in a metropolitan adult population: the Minnesota Heart Survey experience. Am J Public Health. 1984 Apr;74(4):349-52. doi: 10.2105/ajph.74.4.349. PMID 6703162
- [Background] Gillum RF, Folsom AR, Blackburn H. Decline in coronary heart disease mortality. Old questions and new facts. Am J Med. 1984 Jun;76(6):1055-65. doi: 10.1016/0002-9343(84)90857-x. PMID 6375364
- [Background] Rosamond WD, Shahar E, McGovern PG, Sides TL, Luepker RV. Trends in coronary thrombolytic therapy for acute myocardial infarction (the Minnesota Heart Survey Registry, 1990 to 1993). Am J Cardiol. 1996 Aug 1;78(3):271-7. doi: 10.1016/s0002-9149(96)00276-7. PMID 8759803
- [Background] Luepker RV. Current status of cholesterol treatment in the community: the Minnesota Heart Survey. Am J Med. 1997 Feb 17;102(2A):37-42. doi: 10.1016/s0002-9343(97)00466-x. PMID 9217585
- [Background] Arnett DK, Sprafka JM, McGovern PG, Jacobs DR Jr, Shahar E, McCarty M, Luepker RV. Trends in cigarette smoking: the Minnesota Heart Survey, 1980 through 1992. Am J Public Health. 1998 Aug;88(8):1230-3. doi: 10.2105/ajph.88.8.1230. PMID 9702156
- [Background] Smith MA, Shahar E, McGovern PG, Kane RL, Doliszny KM, Arnett DK, Luepker RV. HMO membership and patient age and the use of specialty care for hospitalized patients with acute stroke: The Minnesota Stroke Survey. Med Care. 1999 Dec;37(12):1186-98. doi: 10.1097/00005650-199912000-00002. PMID 10599600
- [Background] Smith MA, Doliszny KM, Shahar E, McGovern PG, Arnett DK, Luepker RV. Delayed hospital arrival for acute stroke: the Minnesota Stroke Survey. Ann Intern Med. 1998 Aug 1;129(3):190-6. doi: 10.7326/0003-4819-129-3-199808010-00005. PMID 9696726
- [Background] Evenson KR, Rosamond WD, Luepker RV. Predictors of outpatient cardiac rehabilitation utilization: the Minnesota Heart Surgery Registry. J Cardiopulm Rehabil. 1998 May-Jun;18(3):192-8. doi: 10.1097/00008483-199805000-00002. PMID 9632320
- [Background] Jacobs DR Jr, Kroenke C, Crow R, Deshpande M, Gu DF, Gatewood L, Blackburn H. PREDICT: A simple risk score for clinical severity and long-term prognosis after hospitalization for acute myocardial infarction or unstable angina: the Minnesota heart survey. Circulation. 1999 Aug 10;100(6):599-607. doi: 10.1161/01.cir.100.6.599. PMID 10441096
- [Background] Phillips EL, Arnett DK, Himes JH, McGovern PG, Blackburn H, Luepker RV. Differences and trends in antioxidant dietary intake in smokers and non-smokers, 1980-1992: the Minnesota Heart Survey. Ann Epidemiol. 2000 Oct;10(7):417-23. doi: 10.1016/s1047-2797(00)00064-8. PMID 11018344
- [Background] Luepker RV, Herlitz J. Differences in the treatment of acute myocardial infarction between regions of countries and the impact on prognosis. J Cardiovasc Risk. 1999 Apr;6(2):77-87. doi: 10.1177/204748739900600204. PMID 10353067
- [Background] McGovern PG, Jacobs DR Jr, Shahar E, Arnett DK, Folsom AR, Blackburn H, Luepker RV. Trends in acute coronary heart disease mortality, morbidity, and medical care from 1985 through 1997: the Minnesota heart survey. Circulation. 2001 Jul 3;104(1):19-24. doi: 10.1161/01.cir.104.1.19. PMID 11435332
- [Background] Vargas A, Doliszny K, Herlitz J, Karlsson T, McGovern P, Brandrup-Wognsen G, Luepker RV. Characteristics and outcomes among patients undergoing coronary artery bypass grafting in western Sweden and Minneapolis-St Paul, Minnesota. Am Heart J. 2001 Dec;142(6):1080-7. doi: 10.1067/mhj.2001.118114. PMID 11717615
- [Background] Arnett DK, McGovern PG, Jacobs DR Jr, Shahar E, Duval S, Blackburn H, Luepker RV. Fifteen-year trends in cardiovascular risk factors (1980-1982 through 1995-1997): the Minnesota Heart Survey. Am J Epidemiol. 2002 Nov 15;156(10):929-35. doi: 10.1093/aje/kwf133. PMID 12419765
- [Background] Barber CA, Margolis K, Luepker RV, Arnett DK. The impact of the Women's Health Initiative on discontinuation of postmenopausal hormone therapy: the Minnesota Heart Survey (2000-2002). J Womens Health (Larchmt). 2004 Nov;13(9):975-85. doi: 10.1089/jwh.2004.13.975. PMID 15665654
- [Background] Crow RS, Hannan PJ, Jacobs DR Jr, Lee SM, Blackburn H, Luepker RV. Eliminating diagnostic drift in the validation of acute in-hospital myocardial infarction--implication for documenting trends across 25 years: the Minnesota Heart Survey. Am J Epidemiol. 2005 Feb 15;161(4):377-88. doi: 10.1093/aje/kwi048. PMID 15692082
- [Background] Arnett DK, Jacobs DR Jr, Luepker RV, Blackburn H, Armstrong C, Claas SA. Twenty-year trends in serum cholesterol, hypercholesterolemia, and cholesterol medication use: the Minnesota Heart Survey, 1980-1982 to 2000-2002. Circulation. 2005 Dec 20;112(25):3884-91. doi: 10.1161/CIRCULATIONAHA.105.549857. Epub 2005 Dec 12. PMID 16344385